CLINICAL TRIAL: NCT00085254
Title: A Safety Run-in/Randomized Phase II Trial of EMD 121974 in Conjunction With Concomitant and Adjuvant Temozolomide With Radiation Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Cilengitide, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02932; NABTT 0306; CDR0000368451; U01CA062475 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-10

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Cilengitide; Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Safety Run In) (Experimental): INITIATION COURSE: Patients receive cilengitide IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  Interventions: Drug: cilengitide; Drug: temozolomide; Radiation: radiation therapy; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase II (Arm1-500mg) (Experimental): INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV (500mg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cilengitide, Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  Interventions: Drug: cilengitide; Drug: temozolomide; Radiation: radiation therapy; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase II (Arm 2 -2000mg) (Experimental): INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV (2000mg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cilengitide,Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  Interventions: Drug: cilengitide; Drug: temozolomide; Radiation: radiation therapy; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Drug: temozolomide — Given orally
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Cilengitide may stop the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving cilengitide together with temozolomide and radiation therapy may kill more tumor cells. This randomized phase I/II trial is studying the side effects and best dose of cilengitide when given together with temozolomide and radiation therapy and to compare how well they work in treating patients with newly diagnosed glioblastoma multiforme

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety profile of EMD 121974 (cilengitide) when administered as a one-hour infusion twice a week concurrently with concomitant and adjuvant temozolomide with radiation therapy for newly diagnosed glioblastoma multiforme. (Safety Run-In)

II. To estimate overall survival in newly diagnosed patients with glioblastoma multiforme treated with EMD 121974 concurrently with concomitant and adjuvant temozolomide with radiation therapy. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate and compare overall survival between a low dose treatment group and a high dose treatment group in newly diagnosed patients with glioblastoma multiforme treated with EMD 121974 concurrently with concomitant and adjuvant temozolomide with radiation therapy. (Phase II)

II. To determine the toxicity of EMD 121974 (cilengitide) when it is administered in conjunction with concomitant and adjuvant temozolomide with radiation therapy in patients with newly diagnosed glioblastoma multiforme. (Phase II)

III. To evaluate the molecular profile of individual patients and correlate molecular expression profiles with clinical outcomes. (Phase II)

IV. To characterize tumor blood volume, tumor blood flow, and permeability ratios using perfusion MR in newly diagnosed glioblastoma multiforme and follow these parameters during treatment with EMD 121974 (cilengitide). (Phase II)

OUTLINE: This is an open-label, multicenter, safety run-in study of cilengitide followed by a randomized phase II study.

Safety Run-In:

INITIATION COURSE: Patients receive cilengitide IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.

MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cilengitide (3 Pre-defined study dose levels are defined as: 500, 1000 and 2000mg). The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity. If no MTD (maximum tolerable dose) is defined through three steps of the dose escalation process, we will pursue the phase II safety/efficacy study with randomized treatment allocation. Patients will be randomized into one of two pre-specified treatment dosage arms, 500mg group or 2000mg group.

PHASE II:

Patients are stratified according to age (50 and under vs over 50), Karnofsky performance score (60%-80% vs 90%-100%), and tumor status (measurable vs nonmeasurable). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive radiotherapy and temozolomide as in safety run-in initiation course and cilengitide at the lower dose as in safety run-in initiation and maintenance courses.

ARM II: Patients receive radiotherapy and temozolomide as in safety run-in initiation course and cilengitide at the higher dose as in safety run-in initiation and maintenance courses.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 9-112 patients (9-18 for safety run-in and 94 [47 per treatment arm] for phase II) will be accrued for this study within 1.5-37 months

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)
* Patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.5 mg/dl or creatinine clearance >= 60 mL/min
* Total bilirubin =< 1.5 mg/dl
* Transaminases =< 4 times above the upper limits of the institutional normal
* Patients must be able to provide written informed consent
* Patients must have recovered from the immediate post-operative period and be maintained on a stable corticosteroid regimen (no increase for 5 days) prior to the start of treatment
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; women of childbearing potential must have a negative pregnancy test
* Patients must have a Mini Mental State Exam score of >= 15
* Patients must have tumor tissue form completed and signed by a pathologist

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents)
* Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin; patients who have been free of disease (any prior malignancy) for >= five years are eligible for this study
* Patients who are unable to undergo an MRI evaluation
* Patients with a history of wound-healing disorders, advanced coronary disease, or with a recent history (# 1 year) of peptic ulcer disease are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Nabors, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Nabors LB, Mikkelsen T, Hegi ME, Ye X, Batchelor T, Lesser G, Peereboom D, Rosenfeld MR, Olsen J, Brem S, Fisher JD, Grossman SA; New Approaches to Brain Tumor Therapy (NABTT) Central Nervous System Consortium. A safety run-in and randomized phase 2 study of cilengitide combined with chemoradiation for newly diagnosed glioblastoma (NABTT 0306). Cancer. 2012 Nov 15;118(22):5601-7. doi: 10.1002/cncr.27585. Epub 2012 Apr 19. PMID 22517399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study sponsored by CTEP and conducted by New Approaches to Brain Tumor Therapy (NABTT). Pts accrued between April 2005 and December 2007. Pts were accrued from 11 Cancer Centers nation wide, in an outpatient setting. All pts had undergone previous surgery and had diagnosis of glioblastoma
Groups:
- Arm 1 (Safety Run In): INITIATION COURSE: Patients receive cilengitide IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 2 - Phase II (Treatment 1): INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV (500mg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cilengitide, Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 3 - Phase II (Treatment 2): INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV (2000mg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cilengitide,Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Arm 1 (Safety Run In) | Arm 2 - Phase II (Treatment 1) | Arm 3 - Phase II (Treatment 2)
Started | 18 | 46 | 48
Completed | 18 | 46 | 48
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: pt had undergone previous surgery and had histological diagnosis of glioblastoma. All pt 18 years or older and KPS greater or equal to 60%
Groups:
- Arm 1 - Safety Run In: INITIATION COURSE: Patients receive cilengitide IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 2 - Phase 2 (Treatment 1): INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (500mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 3 - Phase 2 (Treatment 2): INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (2000mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Safety Run In | Arm 2 - Phase 2 (Treatment 1) | Arm 3 - Phase 2 (Treatment 2) | Total
Number analyzed (Participants) | 18 | 46 | 48 | 112
Age, Continuous [Median (Full Range); unit: years] | 55.6 [22 to 88] | 56.3 [35 to 88] | 54.9 [22 to 81] | 55.5 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 18 | 19 | 46
  Male | 9 | 28 | 29 | 66
Karnofsky Performance Status [Number; unit: participants] — 100 - Normal; no complaints; no evidence of disease 90 - Able to carry on normal activity; minor signs or symptoms of disease 80 - Normal activity with effort; some signs or symptoms of disease 70 - Cares for self; unable to carry on normal activity or to do active work 60 - Requires occasional assistance, but is able to care for most of his personal needs
  participants
    100 | 4 | 8 | 15 | 27
    90 | 6 | 27 | 18 | 51
    80 | 5 | 3 | 7 | 15
    70 | 3 | 6 | 6 | 15
    60 | 0 | 2 | 2 | 4
Surgical Proceedure [Number; unit: participants]
  biopsy | 6 | 10 | 9 | 25
  craniotomy | 12 | 35 | 39 | 86
  other | 0 | 1 | 0 | 1
Corticosteroid Therapy [Number; unit: participants]
  Yes | 13 | 33 | 36 | 82
  No | 4 | 13 | 11 | 28
  missing data | 1 | 0 | 1 | 2
MGMT Statis [Number; unit: participants] — 0-6-methylguanine-DNA methyltransferase
  participants
    methylated | 3 | 11 | 7 | 21
    unmethylated | 9 | 21 | 18 | 48
    unknown | 6 | 14 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities of EMD + RT and TMZ
Description: pts will be evaluated from first dose through end of initiation cycle. (6 weeks of RT+TMZ +EMD and 4 weeks of EMD alone) to review dose limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I)
  DLT defined as: Known TMZ hematological toxicities will not be considered dose limiting.
  Nonhematological toxicities Grades 3-4 severity (except nausea and vomiting without sufficient antiemetic prophylaxis)
Time Frame: 10 weeks
Population: at least 3 pts per cohort will be used to review DLT rate for dose escalation in stepwise fashion. we will enroll 6 pts to ensure that 3 pts are evaluable due to high drop out rate.
Measure: Number; unit: participants
Groups:
- Arm 1 500mg (Safety Run In): INITIATION COURSE: Patients receive cilengitide 500 mg IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  Doses of cilengitide: 500mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  DLT defined as: Known TMZ hematological toxicities will not be considered dose limiting.
  Nonhematological toxicities Grades 3-4 severity (except nausea and vomiting without sufficient antiemetic prophylaxis)
- ARM 2 1000mg (Safety run-in): INITIATION COURSE: Patients receive cilengitide 1000 mg IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  Doses of cilengitide: 1000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  DLT defined as: Known TMZ hematological toxicities will not be considered dose limiting.
  Nonhematological toxicities Grades 3-4 severity (except nausea and vomiting without sufficient antiemetic prophylaxis)
- Arm 3 2000mg (Safety Run-In): INITIATION COURSE: Patients receive cilengitide 2000 mg IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  Doses of cilengitide: 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  DLT defined as: Known TMZ hematological toxicities will not be considered dose limiting.
  Nonhematological toxicities Grades 3-4 severity (except nausea and vomiting without sufficient antiemetic prophylaxis)
Arm/Group | Arm 1 500mg (Safety Run In) | ARM 2 1000mg (Safety run-in) | Arm 3 2000mg (Safety Run-In)
Number analyzed (Participants) | 3 | 4 | 6
participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated or Tolerable Dose (MTD) - 3 Pre-defined Doses
Description: pts will be evaluated from first dose through end of initiation cycle. (6 weeks of RT+TMZ +EMD and 4 weeks of EMD alone) to review any dose limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (safety run-in)
  DLT defined as: Known TMZ hematological toxicities will not be considered dose limiting.
  cohorts at these 3 defined doses: 500mg, 1000mg and 2000mg MTD defined as: dose producing DLT in 2 out of 6 patients or dose level below the dose which produced DLT in >/= 2 out of 3 patients, or in >/= 3 out of 6 patients If no MTD (maximum tolerable dose) was defined through 3 steps of dose escalation, phase 2 will proceed with a randomized treatment allocation of the two pre-specified dosage arms: low dose; 500mg and high dose; 2000mg
Time Frame: 10 weeks
Population: at least 3 pts per cohort will be used to review MTD rate for dose escalation in stepwise fashion of 3 defined doses: 500, 1000 and 2000mg. We will enroll 6 pts to ensure that 3 pts are evaluable due to high drop out rate.
Measure: Number; unit: mg
Arm/Group | Arm 1 - Safety Run In
Number analyzed (Participants) | 13
mg | NA — MTD not achieved. No DLTs at any dose level that were sufficient to define a maximum tolerated dose. Toxicities were equally distributed across all 3 dose levels.

3. Secondary Outcome: Overall Survival Based on Dose Level - Phase 2
Description: survival calculated from date of initial histologic diagnosis and occurence of death. Pts at 500mg dose compared against Pts treated at 2000mg dose. Calculated using median
Time Frame: Up to 3 years
Population: Phase 2 subjects only - does not include the 18 subjects from the safety run-in portion of study
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1 - Phase 2 (Treatment 1): INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (500mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 2 - Phase 2 (Treatment 2): INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (2000mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Arm 1 - Phase 2 (Treatment 1) | Arm 2 - Phase 2 (Treatment 2)
Number analyzed (Participants) | 46 | 48
months | 17.4 [13.3 to 21.6] | 20.8 [7 to 24]
Statistical Analysis 1: Comparison: Arm 1 - Phase 2 (Treatment 1) vs Arm 2 - Phase 2 (Treatment 2); Test type: Superiority or Other; p = 0.4, Regression, Cox; Hazard Ratio (HR) = .83, 95% CI 2-sided [0.5 to 1.3]

4. Secondary Outcome: Frequency of Hematologic and Nonhematologic Adverse Events
Description: The proportion of patients with grade 3 and grade 4 hematologic and non hematologic adverse events per CTCAE 4.0
Time Frame: Up to 1 year
Measure: Number; unit: Number of grade 3 or 4 events
Groups:
- Arm 1- Phase 2 (500mg): INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (500mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm 2 - Phase 2 (2000mg): INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (2000mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Arm 1- Phase 2 (500mg) | Arm 2 - Phase 2 (2000mg)
Number analyzed (Participants) | 46 | 48
Number of grade 3 or 4 events | 48 | 35

5. Primary Outcome: Overall Survival (Phase II)
Description: The overall survival is calculated from time of histological diagnosis to death occurance - median based on all 112 patients, all dose levels
Time Frame: up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 4 (Overall Study): INITIATION COURSE: Patients receive cilengitide IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Arm 4 (Overall Study)
Number analyzed (Participants) | 112
months | 19.7 [16.6 to 21.9]
Statistical Analysis 1: Comparison: Arm 4 (Overall Study); Primary endpoint death - defined from histological diagnosis to death. we assume pt in the study will have overall failure rate of 0.56 per person-year of f/up, a 30% reduction compared to hazard rate of 0.8 per person-year in historical NABTT database. Expected hazard ratio is 0.7 and cohort will produce 63 events among total of 94 pt planned f/up. One-sided test, have 95% power to detect observed ratio of 0.7 at alpha level of 0.1, or we have 88% power at alpha of 0.5 statistical significant; Test type: Superiority or Other; p = 0.0001, Log Rank — adjusted for age: p=.0003, kps: p=.004; and surgical procedure: p=.003; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.3 to 0.5]

ADVERSE EVENTS:
Time Frame: From first dose of treatment in initiation phase until patient progresses on treatment, last dose, off treatment.
Groups:
- Dose 500: INITIATION COURSE: Patients receive cilengitide (500mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (500mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Dose 1000: INITIATION COURSE: Patients receive cilengitide (1000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (2000mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Dose 2000: INITIATION COURSE: Patients receive cilengitide (2000mg) IV over 1 hour on days 1 and 4. Treatment repeats weekly for 10 weeks. Patients also receive oral temozolomide and undergo radiotherapy one hour later on days 1-5 of weeks 1-6.
  MAINTENANCE COURSES: Patients receive oral temozolomide once daily on days 1-5 in courses 1-6. Patients also receive cilengitide (2000mg) IV on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Doses of cilengitide: 500mg, 1000mg and 2000mg
  Temozolimide, Radiation Therapy, laboratory biomarker analysis, pharmacological study
  cilengitide: Given IV
  temozolomide: Given orally
  radiation therapy: Undergo radiotherapy
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Dose 500 | Dose 1000 | Dose 2000
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/6 | 1/54
Other Adverse Events (participants affected / at risk) | 11/52 | 0/6 | 14/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 500 (N=52) | Dose 1000 (N=6) | Dose 2000 (N=54)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema Face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 500 (N=52) | Dose 1000 (N=6) | Dose 2000 (N=54)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) — thrombosis
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
blood -other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study is safety run-in / phase 2 study. Pre-defined doses in safety run-in, 500, 1000 & 2000mg. Safety run-in is under an assumption of low probability of DLT with these dosages. NO actual MTD was defined in the safety run in, all doses were safe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less